CLINICAL TRIAL: NCT02810522
Title: A Registration Study to Assess User Performance of OneTouch Select® Plus Blood Glucose Monitoring System
Brief Title: OneTouch Select® [Brand Name]Plus Blood Glucose Monitoring System(BGMS) Registration Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Medical, China (Industry)
Collaborators: Shanghai 6th People's Hospital (Other); Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Diagnostic
Other Study IDs: LFS-201601
Record Dates: First submitted 2016-06-08; First posted 2016-06-23 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Blood Glucose Measurement

INTERVENTIONS:
Device: OneTouch Select® Plus Glucose Test Strips

SUMMARY:
This study is to support the regulatory application of OneTouch Select® Plus test strips in China. The blood glucose test strip is regulated as an In Vitro Diagnostic (IVD) product and China Food and Drug Administration (CFDA) regulation of IVDs should be complied with. The result of this study will be used to support regulatory filing in China.

Investigational Product:

OneTouch Select® Plus test strips (test with OneTouch Select® Plus glucose meter)

Objectives:

1. Assess Lay User and Health Care Professional (HCP) fingertip test results obtained on OneTouch Select® Plus BGMS compared to a validated method (YSI 2300 glucose analyzer results), according to International Standards Organization( ISO) 15197:2003(E) section 8.0 and ISO 15197:2013(E)
2. Lay User System Use evaluation.
3. Assess the effectiveness of the instructions for use of OneTouch Select® Plus BGMS (Owner's booklet) and insert of test strips for the lay user.

Comparator(control) Product:

YSI 2300 glucose analyser

Acceptance Criteria:

User Performance of the OneTouch Select® Plus Blood Glucose Monitoring system(described as OneTouch Select Plus below) is met if the lay user and HCP results obtained with OneTouch Select Plus meet the requirement stated in section 7.4.1 of ISO () 15197:2003(E). Further to meet the requirements of ISO 15197:2013(E) , the lay user results obtained with OneTouch Select Plus should meet the requirements stated in section 8.2 of ISO 15197:2013(E). The effectiveness of instructions for use is met , if for each item on the Instructions for Use Questionnaire, the 90% lower confidence limit (90% LCL) for the correct response rate is equal to or greater than 70%.

Study Design and subject population:

This study is an open, non-randomized clinical evaluation and will be conducted at a minimum of 2 sites in China. At least 240 evaluable diabetic subjects who meet the enrolment criteria will participate in this evaluation.

Study procedures:

1. Each potential Subject (or legally authorized representative) reads and signs the Informed Consent Form, and receives a signed copy.
2. After completing an in-clinic familiarization session, the Subject lances a fingertip, obtains a drop of blood large enough for two meter tests, and performs a self-test using OneTouch Select Plus BGMS.
3. Study staff immediately performs a blood glucose test from the same blood drop with a second set of OneTouch Select Plus BGMS with the same lot of test strips.
4. Within 5 minutes of the Subject's self-lancing, study staff collects blood from the same finger puncture for hematocrit and reference plasma glucose testing (duplicate tests on the YSI 2300 performed by study staff).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. Subject has a current diagnosis of type 1 or type 2 diabetes mellitus.
3. Subject is currently performing unassisted self-monitoring of blood glucose.
4. Subject agrees to sign two (2) copies each of the Subject Informed Consent Form.
5. Subject agrees to provide relevant demographic, medical history and diabetes management information and agrees to allow study staff access to medical records when necessary.
6. Subject can read and understand Chinese.
7. Subject agrees to complete all aspects of the study including at least one fingertip puncture, one retry in maximum may be performed if insufficient blood collected or an error message is obtained on the first attempt.

Exclusion Criteria:

1. Subject is currently working for, has previously worked for, or has an immediate family member working for a company manufacturing and/or marketing blood glucose monitoring products.
2. Subject has already participated in this study.
3. Subject is knowingly pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2016-11-30 (Estimated); Study Completion 2017-03-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of glucose results obtained from OneTouch Select Plus BGMS | instantly after Glucose testing
  User Performance of the OneTouch Select® Plus Blood Glucose Monitoring system(described as OneTouch Select Plus below) is met if the lay user and HCP results obtained with OneTouch Select Plus meet the requirement stated in section 7.4.1 of ISO 15197:2003(E).Further to meet the requirements of ISO 15197:2013(E) , the lay user results obtained with OneTouch Select Plus should meet the requirements stated in section 8.2 of ISO 15197:2013(E).
The correct response rate of Instructions for Use Questionnaire | instantly after Glucose testing
  The effectiveness of instructions for use is met , if for each item on the Instructions for Use Questionnaire, the 90% lower confidence limit (90% LCL) for the correct response rate is equal to or greater than70%